CLINICAL TRIAL: NCT02099240
Title: Prospective Randomized Study to Compare Clinical Outcomes in Patients With Osteomyelitis Treated With Intravenous Antibiotics Versus Intravenous Antibiotics With an Early Switch to Oral Antibiotics
Brief Title: Patients Response to Early Switch To Oral:Osteomyelitis Study
Acronym: PRESTO:Osteo
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not enough patient enrollment and lack of staffing
Sponsor: Julio Ramirez (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Julio Ramirez, Professor of Medicine, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14.0185
Record Dates: First submitted 2014-03-18; First posted 2014-03-28 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; IV Antibiotics; Oral Antibiotics
MeSH Terms: conditions — Osteomyelitis | interventions — Anti-Bacterial Agents; Amoxicillin; Ampicillin; bacampicillin; carbenicillin indanyl; Carbenicillin; Mezlocillin; Piperacillin; Ticarcillin; Amoxicillin-Potassium Clavulanate Combination; sultamicillin; Penicillin G; Cloxacillin; Dicloxacillin; Methicillin; Oxacillin; benzathine; Potassium; Procaine; Penicillin V; Piperacillin, Tazobactam Drug Combination; ticarcillin-clavulanic acid; Nafcillin; Cefaclor; Cefamandole; cefamandole nafate; Cefonicid; Cefotetan; Cefoxitin; Cefprozil; Cefmetazole; Cefuroxime; cefuroxime axetil; loracarbef; Cefdinir; Ceftibuten; Cefoperazone; Cefixime; Cefotaxime; Cefpodoxime Proxetil; Ceftazidime; Ceftizoxime; Ceftriaxone; Cefepime; Azithromycin; Clarithromycin; Clindamycin; dirithromycin; Erythromycin; benzoyl peroxide, erythromycin drug combination; Lincomycin; Cinoxacin; Ciprofloxacin; Enoxacin; Gatifloxacin; grepafloxacin; Levofloxacin; lomefloxacin; Moxifloxacin; Nalidixic Acid; Norfloxacin; Ofloxacin; sparfloxacin; Cilastatin, Imipenem Drug Combination; Meropenem; Aztreonam; Amikacin; Gentamicins; Kanamycin; Neomycin; Netilmicin; Streptomycin; Tobramycin; Paromomycin; Vancomycin; Demeclocycline; Doxycycline; Methacycline; Minocycline; Oxytetracycline; Tetracycline; Chlortetracycline; Mafenide; Silver Sulfadiazine; Sulfacetamide; Sulfadiazine; Sulfamethoxazole; Sulfasalazine; Sulfisoxazole; Trimethoprim, Sulfamethoxazole Drug Combination; Thymidine Monophosphate; Sulfamethizole; Rifabutin; Rifampin; rifapentine; Linezolid; quinupristin-dalfopristin; Bacitracin; Chloramphenicol; Fosfomycin; Isoniazid; Methenamine; methenamine hippurate; methenamine mandelate; Benchmarking; Metronidazole; Mupirocin; Nitrofurantoin; Nitrofurazone; Novobiocin; Polymyxin B; Spectinomycin; Trimethoprim; Colistin; Cycloserine; Capreomycin; Ethionamide; Pyrazinamide; Erythromycin Ethylsuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous antibiotics (Active Comparator): Intravenous antibiotics for the full duration of therapy
  Interventions: Procedure: intravenous antibiotics
- oral antibiotics (Active Comparator): intravenous antibiotic therapy plus early switch to oral antibiotic therapy
  Interventions: Drug: oral antibiotics

INTERVENTIONS:
Drug: oral antibiotics — intravenous antibiotics with early switch to oral antibiotics, antibiotic type will be dependent on bacteria type
  Other Names: Amoxicillin; Amoxil®; Ampicillin; Omnipen®; Bacampicillin; Spectrobid®; Carbenicillin Indanyl; Pyopen®, Geogen®, Geocillin®; Mezlocillin; Mezlin®; Piperacillin*; Pipracil®; Ticarcillin; Ticar®; Amoxicillin-Clavulanic Acid; Augmentin®; Ampicillin-Sulbactam*; Unasyn®; Benzylpenicillin; Benpen®; Cloxacillin; Tegopen®, Coxapen®; Dicloxacillin; Dycill®, Dynapen®, Pathocil®; Methicillin; Staphcillin®; Oxacillin; Prostaphilin®, Bactocil®; Penicillin G (Benzathine, Potassium, Procaine); Bicillin® C-R/L-A, Pfizerpen®, Wycellin®; Penicillin V; Pen-Veek®, Beepen-VK®; Piperacillin+Tazobactam*; Zozyn®; Ticarcillin+Clavulanic Acid; Timentin®; Nafcillin; Unipen®, Nafcil®; Cefaclor; Ceclor®, Ceclor CD®; Cefamandol; Mandol®; Cefonicid; Monocid®; Cefotetan; Cefotan®; Cefoxitin; Mefoxin®; Cefprozil; Cefzil®; Ceftmetazole; Zefazone®; Cefuroxime; Kefurox®, Zinacef®; Cefuroxime axetil; Ceftin®; Loracarbef; Lorabid®Cefdinir; Omnicef®; Ceftibuten; Cedax®; Cefoperazone; Cefobid®; Cefixime*; Suprax®; Cefotaxime*; Claforan®; Cefpodoxime proxetil; Vantin®; Ceftazidime*; Ceptaz®, Fortaz®, Tanicef®; Ceftizoxime*; Cefizox®; Ceftriaxone*; Rocephin®; Cefepime; Maxipime®; Azithromycin*; Zithromax®; Clarithromycin*; Biaxin®; Clindamycin; Cleocin®; Dirithromycin; Dynabac®; Erythromycin; E-mycin®, Ery-tab®, Benzamycin®; Lincomycin; Lincocin®; T roleandomycin; T ao®; Cinoxacin; Cinoxacin®; Ciprofloxacin*; Cipro®; Enoxacin; Penetrex®; Gatifloxacin; T equin®; Grepafloxacin; Levofloxacin; Levaquin®, Quixin®; Lomefloxacin; Maxaquin®; Moxifloxacin; A velox®; Nalidixic acid; NegGam®; Norfloxacin*; Noroxin®; Ofloxacin; Floxin®; Sparfloxacin; Zagam®; T rovafloxacin; T rovan®; Imipenem-Cilastatin*; Primaxin®; Meropenem; Merrem®; Aztreonam*; Azactam®; Amikacin*; Amikin®; Gentamicin; Garamycin®; Kanamycin; Kantrex®; Neomycin; Mycifradin®, Neo-Fradin®; Netilmicin; Netromycin®; Streptomycin; Streptomycin®; T obramycin*; Tobrex®, Nebcin®; Paromomycin; Humatin®; T eicoplanin; T argocid®; Vancomycin*; Vancocyn®, Lyphocin®; Demeclocycline; Declomycin®; Doxycycline; Doxy®, Vibra®, Vibramycin®; Methacycline; Rondomycin®; Minocycline; Minocin®; Oxytetracycline; Terramycin®; T etracycline; Sumycin®; Chlortetracycline; Mafenide; Sulfamylon®; Silver Sulfadiazine; SSD®, Silvadene®; Sulfacetamide; Sultrim®; Sulfadiazine; Sulfamethoxazole; Gantanol®; Sulfasalazine; Sulfasalazine®,Azulfidine®; Sulfisoxazole; T rimethoprim-Sulfamethoxazole; Bactrim®, Septra®, Cofatrim®, Primsol®; Sulfamethizole; Thiosulfil Forte®; Rifabutin; Mycobutin®; Rifampin; Rifadin®; Rifapentine; Priftin®; Linezolid*; Zyvox®; Quinopristin+Dalfopristin*; Synercid®; Bacitracin; Baci-IM; Chloramphenicol*; Chloromycetin®; Colistemetate; Coly-Mycin® M & S; Fosfomycin; Monurol®; Isoniazid; Rifamate®; Methenamine; Hiprex®, Mandelamine®; Metronidazol; Flagyl®; Mupirocin; Bactroban®; Nitrofurantoin; Macrobid®, Macrodantin®, Furantoin®; Nitrofurazone; Furacin®; Novobiocin; Albamycin®; Polymyxin B; Aerospin®; Spectinomycin; T robicin®; T rimethoprim; Proloprim®, Trimpex®; Colistin; Cycloserine; Capreomycin; Ethionamide; Pyrazinamide; Para-aminosalicyclic acid; Erythromycin ethylsuccinate + sulfisoxazole
  Arms: oral antibiotics
Procedure: intravenous antibiotics — intravenous antibiotics for the full duration of therapy, antibiotic type will be dependent on bacteria type
  Other Names: Amoxicillin; Amoxil®; Ampicillin; Omnipen®; Bacampicillin; Spectrobid®; Carbenicillin Indanyl; Pyopen®, Geogen®, Geocillin®; Mezlocillin; Mezlin®; Piperacillin*; Pipracil®; Ticarcillin; Ticar®; Amoxicillin-Clavulanic Acid; Augmentin®; Ampicillin-Sulbactam*; Unasyn®; Benzylpenicillin; Benpen®; Cloxacillin; Tegopen®, Coxapen®; Dicloxacillin; Dycill®, Dynapen®, Pathocil®; Methicillin; Staphcillin®; Oxacillin; Prostaphilin®, Bactocil®; Penicillin G (Benzathine, Potassium, Procaine); Bicillin® C-R/L-A, Pfizerpen®, Wycellin®; Penicillin V; Pen-Veek®, Beepen-VK®; Piperacillin+Tazobactam*; Zozyn®; Ticarcillin+Clavulanic Acid; Timentin®; Nafcillin; Unipen®, Nafcil®; Cefaclor; Ceclor®, Ceclor CD®; Cefamandol; Mandol®; Cefonicid; Monocid®; Cefotetan; Cefotan®; Cefoxitin; Mefoxin®; Cefprozil; Cefzil®; Ceftmetazole; Zefazone®; Cefuroxime; Kefurox®, Zinacef®; Cefuroxime axetil; Ceftin®; Loracarbef; Lorabid®Cefdinir; Omnicef®; Ceftibuten; Cedax®; Cefoperazone; Cefobid®; Cefixime*; Suprax®; Cefotaxime*; Claforan®; Cefpodoxime proxetil; Vantin®; Ceftazidime*; Ceptaz®, Fortaz®, Tanicef®; Ceftizoxime*; Cefizox®; Ceftriaxone*; Rocephin®; Cefepime; Maxipime®; Azithromycin*; Zithromax®; Clarithromycin*; Biaxin®; Clindamycin; Cleocin®; Dirithromycin; Dynabac®; Erythromycin; E-mycin®, Ery-tab®, Benzamycin®; Lincomycin; Lincocin®; T roleandomycin; T ao®; Cinoxacin; Cinoxacin®; Ciprofloxacin*; Cipro®; Enoxacin; Penetrex®; Gatifloxacin; T equin®; Grepafloxacin; Levofloxacin; Levaquin®, Quixin®; Lomefloxacin; Maxaquin®; Moxifloxacin; A velox®; Nalidixic acid; NegGam®; Norfloxacin*; Noroxin®; Ofloxacin; Floxin®; Sparfloxacin; Zagam®; T rovafloxacin; T rovan®; Imipenem-Cilastatin*; Primaxin®; Meropenem; Merrem®; Aztreonam*; Azactam®; Amikacin*; Amikin®; Gentamicin; Garamycin®; Kanamycin; Kantrex®; Neomycin; Mycifradin®, Neo-Fradin®; Netilmicin; Netromycin®; Streptomycin; Streptomycin®; T obramycin*; Tobrex®, Nebcin®; Paromomycin; Humatin®; T eicoplanin; T argocid®; Vancomycin*; Vancocyn®, Lyphocin®; Demeclocycline; Declomycin®; Doxycycline; Doxy®, Vibra®, Vibramycin®; Methacycline; Rondomycin®; Minocycline; Minocin®; Oxytetracycline; Terramycin®; T etracycline; Sumycin®; Chlortetracycline; Mafenide; Sulfamylon®; Silver Sulfadiazine; SSD®, Silvadene®; Sulfacetamide; Sultrim®; Sulfadiazine; Sulfamethoxazole; Gantanol®; Sulfasalazine; Sulfasalazine®,Azulfidine®; Sulfisoxazole; T rimethoprim-Sulfamethoxazole; Bactrim®, Septra®, Cofatrim®, Primsol®; Sulfamethizole; Thiosulfil Forte®; Rifabutin; Mycobutin®; Rifampin; Rifadin®; Rifapentine; Priftin®; Linezolid*; Zyvox®; Quinopristin+Dalfopristin*; Synercid®; Bacitracin; Baci-IM; Chloramphenicol*; Chloromycetin®; Colistemetate; Coly-Mycin® M & S; Fosfomycin; Monurol®; Isoniazid; Rifamate®; Methenamine; Hiprex®, Mandelamine®; Metronidazol; Flagyl®; Mupirocin; Bactroban®; Nitrofurantoin; Macrobid®, Macrodantin®, Furantoin®; Nitrofurazone; Furacin®; Novobiocin; Albamycin®; Polymyxin B; Aerospin®; Spectinomycin; T robicin®; T rimethoprim; Proloprim®, Trimpex®; Colistin; Cycloserine; Capreomycin; Ethionamide; Pyrazinamide; Para-aminosalicyclic acid; Erythromycin ethylsuccinate + sulfisoxazole
  Arms: Intravenous antibiotics

SUMMARY:
Based on the current literature, investigators hypothesize that patients with osteomyelitis who are treated with the standard approach of intravenous antibiotics for the full duration of therapy will have the same clinical outcomes as patients treated with the experimental approach of intravenous antibiotics with early switch to oral antibiotics.

The primary objective of this study is to compare patients with osteomyelitis treated with the standard approach of intravenous antibiotics for the full duration of therapy versus patients treated with intravenous antibiotics with an early switch to oral antibiotics in relation to clinical outcomes at 12 months after discontinuation of antibiotic therapy. Secondary objectives of the study include the evaluation of adverse events related to the use of antibiotics as well as the cost of care evaluated from the hospital perspective.

DETAILED DESCRIPTION:
1.1. Background Information Osteomyelitis is a common disease associated with significant morbidity and high cost (1). The treatment of osteomyelitis can be challenging requiring prolonged administration of antibiotics and extensive surgical procedures. Even when the infection is treated, the relapse rate is as high as 20% (2). When a bone is infected, the local multiplication of bacteria produces a local inflammatory response with presence of neutrophils and macrophages with areas of microthrombi and avascular necrosis. If a significant area of avascular necrosis develops, a segment of the bone without any blood supply can become separated and form a sequestrum. Since infection of sequestrum occurs in most patients with osteomyelitis, it is considered that in addition to antibiotic treatment, the patient requires surgical intervention for removal of necrotic bone.

1.2. Scientific Rationale There is agreement regarding the minimal duration of antibiotic therapy for patients with osteomyelitis. Since an infected bone may take 3 to 4 weeks to re--- vascularize, the duration of therapy should be a minimum of 4 to 6 weeks of antibiotics. Because different organisms can cause osteomyelitis, the initial antibiotic therapy during hospitalization should include broad---spectrum antibiotics to cover the most likely organisms. As part of the initial management, a bone biopsy is regularly performed to identify the particular etiologic agent. Once the organism and its antimicrobial susceptibilities are known, the spectrum of antibiotic therapy is narrowed, and the antimicrobial therapy continues with an antibiotic that is targeted according to the susceptibility of the identified pathogen. Targeted antibiotic therapy in patients with osteomyelitis is usually performed after 3 to 5 days of broad spectrum antibiotics, since this is the time required by the microbiology department to generate antimicrobial susceptibilities after the bone biopsy is performed. In regard to the route of antibiotic administration, the standard approach is to use an intravenous antibiotic.

1.3. Potential Risks A potential risk for the use of an early switch to oral antibiotics in patients with osteomyelitis is that the blood level achieved with oral antibiotics may not be high enough to attain clinical resolution of the infection.

1.4. Potential Benefits There are several potential benefits of using oral antibiotics instead of intravenous antibiotics. First, avoiding a peripherally inserted central line eliminates the risk of line infection and line---associated deep vein thrombosis. An early switch to oral antibiotics may also facilitate early hospital discharge. A shorter hospital stay will decrease the risk of hospital---associated complications such as hospital---acquired infections. Further, the patients' quality of life may be better without a central line. Finally, the total cost of therapy will be significantly reduced with oral therapy.

2. Methods 2.1. Trial design & setting This will be a prospective, randomized, unblinded clinical trial to define if the clinical outcomes of patients with osteomyelitis treated with the experimental approach of intravenous antibiotics with an early switch to oral therapy is non---inferior to the current standard approach of intravenous antibiotics for the full duration of therapy.

2.8. Sample Size & Statistical Analysis The null hypothesis for this study will be as follows: H0: πs --- πe ≤ ---Δ Where πs is the proportion of clinical failures in the intravenous therapy only group, πe is the proportion of clinical failures in the intravenous therapy plus early switch to oral therapy group, and Δ is the non---inferiority margin. The alternative hypothesis will be: HA: πs --- πe > ---Δ We expect that there will be a 20% clinical failure rate for the primary outcome in both the intravenous antibiotic therapy group and the intravenous antibiotic therapy plus early switch to oral antibiotic therapy group. The study will be powered at 80% with Δ of 0.1. A total of 396 patients will be needed to obtain a 95% confidence interval for the difference in failure rates between the two groups that has a lower limit above ---Δ. If the lower limit of this 95% confidence interval for the 10 difference in clinical failure rates between the two arms is above -Δ, non---inferiority will be met. Considering that approximately 15% of patients will be lost during study follow---up, a total of 456 patients will be enroll in the trial to obtain the 396 patients necessary for final analyses.

3. Data Quality Management Plan 3.1. Overview of the Clinical and Translational Research Support Center

The University of Louisville Clinical and Translational Research Support Center (CTRSC) will be responsible for data collection, data quality, and data analysis for this project. The CTRSC (http://www.ctrsc.net) is a multi---disciplinary team comprised of professionals in medicine, public health, statistics, and computer science. The team has considerable experience managing and supporting single---site and multi---center clinical research studies. Specifically, members of the CTRSC will be responsible for:

* Study design
* Development of data collection forms
* Development of study manual 11
* Development of electronic Internet base data entry system
* Providing instruction on use of forms and data entry system
* Development of study database
* Tracking subject enrollment
* Overseeing data transmission
* Providing data management
* Handling data validation
* Protecting confidentiality of data
* Performing feasibility evaluation The data quality team leader for this project will be Dr. Robert Kelley with assistance from Dr. Timothy Wiemken and Dr. Paula Peyrani.

The CTRSC has access to the University of Louisville's high---performance computing cluster, which consists of 312 IBM iDatplex nodes each with two Intel Xeon quad--- core processors for 2496 total cores. The cluster is equipped with a variety of statistical and bioinformatics software including SAS, R, Matlab, ClustalW, and Blast, and C, Fortran, Perl, and Python libraries. In addition, the CTRSC has several iMac and IBM---compatible workstations with several data management and analysis packages installed including R, Matlab, SQL Server 2012, SAS, SPSS, Eclipse, Visual Studio .NET 2010, MySQL Server 5.1, Tableau 8.0, and REDCap.

3.2. Purpose of Data Quality Management Plan

The purpose of this data quality management plan is outline the procedures and processes necessary to:

1. Ensure the data collection and data management for the study are conducted in a manner consistent with University of Louisville standards as well as state and federal regulations.
2. Ensure that data collected are accurate and complete when verified against source documents.
3. Provide approaches for early interception and correction of errors in data collection.
4. Identify areas where specific education and training efforts regarding data collection need to be focused.
5. Outline the tools that will be used to monitor and assess data quality.
6. Outline the Data Quality Management Team meeting schedule for this project. 3.3. Data Capture Primary data collection will be performed by a qualified study coordinator(s) who will abstract subject data from the electronic medical record onto a paper case report form. Once the paper case report form is complete, the study coordinator or other designee will enter the data into a secure, web---based clinical data management system.

ELIGIBILITY:
Inclusion Criteria:

* Only adult patients will be invited to participate in this trial (age ≥ 18 years). A patient will be considered a candidate to participate in this trial if the following two inclusion criteria are present:

  1. Isolation of an organism from bone culture that is susceptible to intravenous and oral antibiotics.
  2. Plus at least one of the following:

     * Evidence of local inflammatory response, manifested as local pain, edema, erythema, warmth, or drainage.
     * Evidence of systemic inflammatory response, manifested as fever, elevated C---reactive protein (CRP) level, erythrocyte sedimentation rate (ESR), or white blood cell count.
* *Osteomyelitis---compatible findings on plain radiograph, computed tomography, bone scan, magnetic resonance imaging, or positron emission tomography.

  * Pathology report indicative of osteomyelitis.

Exclusion Criteria:

* A patient will not be considered as a candidate to participate in this study if the study team expects the subject to be non---compliant with the study follow---up clinic visit.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Clinical Failures | 1 month
  Clinical failure will be defined as clinical or laboratory evidence of infection collected from the patient's medical record documents.

SECONDARY OUTCOMES:
Evaluation of adverse events related to the use of antibiotics | 1 month
  Antibiotic---related adverse events will be defined according to the Food and Drug Administration adverse events listed in the package insert of the antibiotic prescribed for each subject.
Cost of care from the hospital perspective | 12 months
  Costs will be calculated from the hospital perspective and will include the costs of the antibiotic therapy, home healthcare (nursing--- and infusion---related), and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: David Seligson, MD, Principal Investigator — University of Louisville; Julio Ramirez, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Result] Lew DP, Waldvogel FA. Osteomyelitis. Lancet. 2004 Jul 24-30;364(9431):369-79. doi: 10.1016/S0140-6736(04)16727-5. PMID 15276398
- [Result] Haas DW, McAndrew MP. Bacterial osteomyelitis in adults: evolving considerations in diagnosis and treatment. Am J Med. 1996 Nov;101(5):550-61. doi: 10.1016/s0002-9343(96)00260-4. PMID 8948280
- [Result] Waldvogel FA, Medoff G, Swartz MN. Osteomyelitis: a review of clinical features, therapeutic considerations and unusual aspects. N Engl J Med. 1970 Jan 22;282(4):198-206. doi: 10.1056/NEJM197001222820406. No abstract available. PMID 4902833
- [Result] Lazzarini L, Lipsky BA, Mader JT. Antibiotic treatment of osteomyelitis: what have we learned from 30 years of clinical trials? Int J Infect Dis. 2005 May;9(3):127-38. doi: 10.1016/j.ijid.2004.09.009. PMID 15840453
- [Result] Conterno LO, da Silva Filho CR. Antibiotics for treating chronic osteomyelitis in adults. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD004439. doi: 10.1002/14651858.CD004439.pub2. PMID 19588358
- [Result] Peyrani P, Allen M, Seligson D, Roberts C, Chen A, Haque N, Zervos M, Wiemken T, Harting J, Christensen D, Ramirez R. Clinical outcomes of osteomyelitis patients infected with methicillin-resistant Staphylococcus aureus USA-300 strains. Am J Orthop (Belle Mead NJ). 2012 Mar;41(3):117-22. PMID 22530208